CLINICAL TRIAL: NCT04791774
Title: Systemic Bioavailability of Enteral Protein-bound Versus Free Amino Acid Nutrition During Intestinal Malabsorption in Critical Illness
Brief Title: Protein-bound Versus Free Amino Acid Nutrition During INtestinal Malabsorption in Critical Illness
Acronym: PANINI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL60452.068.17
Record Dates: First submitted 2017-05-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Intestinal Malabsorption; Critical Illness; Protein Malnutrition
Keywords: Proteins; Stable Isotopes; Enteral Nutrition
MeSH Terms: conditions — Malabsorption Syndromes; Critical Illness; Kwashiorkor | interventions — Milk Proteins; Proteins; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein group (Active Comparator): Patients receive 20 grams of Intrinsically labelled milk protein.
  Interventions: Dietary Supplement: Milk protein (food grade protein)
- Free amino acid group (Experimental): Patients receive 20 grams of free amino acids equivalent to the milk protein labelled with 13C-Phenylalanine
  Interventions: Dietary Supplement: Fee amino acids (food grade amino acids)

INTERVENTIONS:
Dietary Supplement: Milk protein (food grade protein) — Subjects will receive an enteral nutritional formula containing 20 grams intrinsically labeled (1-[13C]-phenylalanine) milk protein
  Other Names: Protein
  Arms: Protein group
Dietary Supplement: Fee amino acids (food grade amino acids) — Nutritional formula containing 20 grams of a free amino acid mixture equivalent in composition to the milk protein with 1-[13C]-labeled phenylalanine
  Other Names: Amino Acids
  Arms: Free amino acid group

SUMMARY:
In the current study, we willquantitate the difference in digestion and absorption kinetics of dietary whole protein versus free amino acids in vivo in critically ill patients admitted to the intensive care unit suffering from malabsorption. 16 adult, mechanically ventilated ICU patients with clinical signs of malabsorption (faecal weight >350 g/day) will be included. All patients will receive a primed continuous intravenous infusion of L-[ring2H5]-phenylalanine and L-[3,5-2H2]-Tyrosine for the duration of the study period. After reaching an isotopic steady state (1.5 hours), patients will receive either [1-13C]- phenylalanine labelled milk protein or free amino acids with an identical constitution and [1-13C]-phenylalanine.

Main study endpoint will be the splanchnic extraction of phenylalanine, calculated from systemic [1-13C]- and L-[ring2H5]-phenylalanine enrichment.

DETAILED DESCRIPTION:
Background of the study:

The importance of the provision of sufficient protein in critical illness is increasingly recognized. Protein malabsorption seems to be an underestimated but substantial problem in critically ill patients, limiting the amount of this important nutrient that actually becomes available within the systemic circulation. Among several contributors to malabsorption in critical illness, exocrine pancreatic insufficiency has recently emerged as a regularly occurring phenomenon during critical illness. Pancreatic insufficiency could lead to reduced digestion and subsequent uptake of enteral provided proteins. A proposed solution to this problem could be the use of elementary feeds containing free amino acids instead of whole protein. Due to the lack of easy applicable and reproducible tests for protein malabsorption the true efficacy of these feeds is still unknown. We hypothesize that enteral nutrition containing free amino acids leads to higher systemic levels of amino acids and will therefore increase the amount of dietary amino acids available for protein synthesis.

Objective of the study:

To quantitate the difference in digestion and absorption kinetics of dietary whole protein versus free amino acids in vivo in patients admitted to the ICU suffering from malabsorption.

Study design:

Randomized, single-blind controlled, single-centre, intervention study.

Study population:

16 adult, mechanically ventilated ICU patients with clinical signs of malabsorption (faecal weight >350 g/day).

Intervention:

Normal enteral nutrition will be ceased 8 hours before the start of study participation. All patients will receive a primed continuous intravenous infusion of L-[ring2H5]-phenylalanine and L-[3,5-2H2]-Tyrosine for the duration of the study period. After reaching an isotopic steady state (1.5 hours), patients will receive either [1-13C]- phenylalanine labelled milk protein or free amino acids with an identical constitution and [1-13C]-phenylalanine.

Primary study parameters/outcome of the study:

Main study endpoint will be the splanchnic extraction of phenylalanine, calculated from systemic [1-13C]- and L-[ring2H5]-phenylalanine enrichment.

Secundary study parameters/outcome of the study:

Secondary endpoints include the impact of enteral nutrition on whole body protein balance, glucose and insulin concentrations and faecal energy and protein loss as a measure of malabsorption.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Total study participation will take 16 hours, including 8 hours of fasting. Arterial blood samples will be collected regularly, with 50 ml of blood being sampled in total, amounting to a maximum of 1.0% of total circulating volume. All infusions, as well as blood sample collection, will be performed through indwelling catheters necessary for normal ICU treatment, meaning no lines or nasogastric tubes will have to be placed for the purposes of the study. Both isotopically labelled protein and free amino acids have been proven safe for use in humans and carry no harmful risks for the study participant. Changes in protein digestion, absorption and metabolism are specific to critical illness and their impact on the clinical condition and recovery of patients is severe. Investigating new strategies to modulate these effects are therefore essential, but require experimental studies in a vulnerable population. The risks in the present study are minimal whereas the results could help improve nutritional management in the intensive care.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 75 years
2. Fecal weight > 350g/day
3. Critical illness of any origin (e.g. medical, surgical, trauma) requiring admittance on ICU ward.
4. Expected ICU stay for the duration of the study protocol
5. Mechanically ventilated (PaO2/FiO2 ratio of >100 and <300)
6. Nasogastric tube in situ
7. Receiving full enteral nutrition without gastric residual volumes
8. Arterial (any location) line in situ
9. Flexi-seal system in situ

Exclusion Criteria:

1. Proven (pre-existing) intestinal disease that potentially limits normal gut function and absorption of nutrients (e.g. IBD, short-bowel, entero-cutaneous fistulas including a surgical enterostomy)
2. Proven (pre-existing) primary pancreatic disease or obstruction of the pancreatic duct of any origin (e.g. pancreatitis, carcinoma).
3. Patients who are moribund (not expected to be in ICU for more than 48 hours due to imminent death)
4. A lack of commitment to full aggressive care during the first week due to severity of illness, comorbidities and potential harm from maximal treatment (anticipated withholding or withdrawing treatments)
5. Absolute contraindication to enteral nutrients (e.g., gastrointestinal [GI] perforation, obstruction or no GI tract access for any reason)
6. Receiving parenteral nutrition.
7. Nasoduodenal or nasojejunal feeding tube
8. Renal dysfunction defined as a serum creatinine >171 umol/L or a urine output of less than 500 ml/last 24 hours
9. Patients requiring chronic veno-venous hemofiltration
10. Patients on ECMO/ELS
11. Cirrhosis - Child Pugh class C/D liver disease
12. Patients with primary admission diagnosis of burns (>30% body surface area)
13. Weight less than 50 kg or greater than 100 kg
14. Pregnant patients or lactating with the intent to breastfeed
15. Previous randomization in this study
16. Enrolment in any other interventional study
17. Milk/lactose allergy
18. Previous participation in a 13C amino acid tracer study within the last year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
systemic availability of diet-derived amino acids | 8 hours
  The main study endpoint in this study is the systemic availability of enteral administered protein-bound or free amino acid nutrition, including the rate of appearance (Ra) of dietary derived phenylalanine. Modified Steele's equations will be applied to plasma enrichments of L-[ring-2H5]-phenylalanine, L-[1-13C]-phenylalanine enrichment, L-[ring-2H4]-tyrosine and L-[3,5-2H2]-tyrosine.

SECONDARY OUTCOMES:
Total plasma amino acids (AAmax [μmol/L]) | 8 hours
  Total plasma amino acids (AAmax [μmol/L])
Plasma glucose (glucosemax [mmol/L]) | 8 hours
  Plasma glucose (glucosemax [mmol/L])
Plasma insulin (insulinmax [mU/L]) | 8 hours
  Plasma insulin (insulinmax [mU/L])
Intestinal absorption capacity (energy provided - fecal energy loss x 100%) | 2 x 24 hours
  Intestinal absorption capacity (energy provided - fecal energy loss x 100%)
Fecal elastase (µg elastase / g feces) | 2 x 24 hours
  Fecal elastase (µg elastase / g feces)
Fecal presence of L-[1-13C]-phenylalanine | 2x 12 hours
  Fecal presence of L-[1-13C]-phenylalanine

CONTACTS AND LOCATIONS:
Overall Officials: Marcel van de Poll, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht UMC+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Gassel RJ, Weijzen ME, Kouw IW, Senden JM, Wodzig WK, Olde Damink SW, van de Poll MC, van Loon LJ. Administration of Free Amino Acids Improves Exogenous Amino Acid Availability when Compared with Intact Protein in Critically Ill Patients: A Randomized Controlled Study. J Nutr. 2024 Feb;154(2):554-564. doi: 10.1016/j.tjnut.2023.12.015. Epub 2023 Dec 15. PMID 38103646